CLINICAL TRIAL: NCT05478291
Title: Effect of Vitamin D Supplementation on Surrogate Markers of Atherosclerosis in North Indian Individuals With Pre-diabetes and Low Vitamin D Levels: a Randomised Controlled Trial.
Brief Title: Vitamin D Supplementation on Surrogate Markers of Atherosclerosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diabetes Foundation, India (Other)
Responsible Party: Principal Investigator, Dr Anoop Misra, President, Diabetes Foundation, India
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2021-8753
Record Dates: First submitted 2022-04-27; First posted 2022-07-28 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Atherosclerosis
Keywords: Vitamin D; Prediabetes; Asian Indians
MeSH Terms: conditions — Atherosclerosis; Prediabetic State

STUDY DESIGN:
Intervention Model Description: A randomized open labelled placebo-controlled trial.
Masking Description: Both participants and their clinical care team will be aware of the allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vitamin D supplementation (Experimental): Appropriate diet and physical activity counselling
  Supplementation with Vitamin D and oral Calcium- Doses of cholecalciferol (commercial name, Calcirol) 60,000 international units (sachets, dissolved in half glass milk) once per week for eight weeks to intervention group and placebo (Lactose granules) to the placebo group according to the random numbers generated by the computer.
  After every 24 weeks blood 25 (OH) D levels will be assessed. If the subjects are found to be still deficient then supplementation of cholecalciferol 60,000 IU per week for eight weeks will be repeated. If the 25 (OH) D levels are normal, then cholecalciferol supplementation in doses of 200 international units per day will be given as a maintenance dose.
  Interventions: Other: Vitamin D supplementation

INTERVENTIONS:
Other: Vitamin D supplementation — Appropriate diet and physical activity counselling to both groups. Supplementation with Vitamin D and oral Calcium-Doses of cholecalciferol (commercial name, Calcirol) 60,000 IU (sachets, dissolved in half glass milk) once per week for eight weeks for the intervention group and placebo (Lactose granules) to the placebo group according to the random numbers generated by the computer. After every 24 weeks blood 25 (OH) D levels will be assessed. If the subjects are found to be still deficient then supplementation of cholecalciferol 60,000 IU per week for eight weeks will be repeated.If the 25 (OH) D levels are normal, then cholecalciferol supplementation in doses of 200 IU per day will be given as a maintenance dose. Equal doses of calcium carbonate (1gm per day, commercial name Calcal) will be given to both the groups.

SUMMARY:
For this study, our sample population is individuals with prediabetes, who are at an increased risk for atherosclerosis. In this proposed randomized placebo-controlled prospective trial, we would be enrolling 120 subjects with prediabetes having vitamin D deficiency. These subjects will be randomized into two groups; lifestyle modification counselling along with intervention with either vitamin D supplementation or placebo. Clinical and dietary profiles including sunlight exposure, anthropometry, glycemic and lipid profiles, fasting insulin, adiponectin, body composition (DEXA), skinfolds (4 sites), surrogate markers of atherosclerosis/inflammation (TNF-alpha, hs-CRP, Matrix Metalloproteinase-9, flow-mediated dilatation of brachial artery, pulse wave velocity, and carotid intima-mediated thickness) will be measured at week 0 and week.

DETAILED DESCRIPTION:
Prediabetes is a substantial problem in India not only because it itself can be associated with morbidities such as coronary artery disease but also because it is a point of important for prevention of diabetes. It is not clear if vitamin D supplementation in Indian population associated with heightened tendency for prediabetes, metabolic syndrome, atherosclerosis and dys-metabolic state etc. could, besides lifestyle factors, be related to vitamin D deficiency, or interaction between the two. This study is based on the assumption that the supplementation of vitamin D may decrease Atherosclerosis in individuals with prediabetes.

Supplementation of vitamin D is of major significance in terms of economic and health benefits to the individual and to the country. In addition, such simple and low-cost measures would help maintain a normal metabolic system. The proposed study would also lead to a community-based model of education regarding metabolic and cardiovascular disease. This study will help to develop slandered protocol for the prevention and treatment of non-communicable diseases (NCDs).

In India, the prevalence of coronary heart disease (7%-13% in urban and 2%-7% in rural populations), as well as diabetes, is high. Positive results from this study may benefit a large number of individuals at risk for cardiovascular disease. In addition, If vitamin D supplementation leads to decreased atherosclerosis as indicated by surrogate markers of atherosclerosis, it may be a cost-effective and novel way to reduce or prevent atherosclerosis in the Indian population, which is at high risk for the development of atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Pre-diabetes: fasting blood glucose ≥100mg/dl and <125.99mg/dl, 2-h plasma glucose ≥140mg/dl and <200mg/dl (after ingestion of 75 g anhydrous oral glucose).
* Baseline level of 25 hydroxy vitamin D <30ng/dl and aged 20-60 years.

Exclusion Criteria:

* Received Vitamin D and/or calcium supplementation in the previous six months, on any medication within the last one month which could potentially influence insulin secretion, insulin sensitivity, vitamin D or calcium metabolism (eg metformin, thiazolidione, steroids etc) and on any medication that activate steroid and xenobiotic receptor and drugs used in transplantation (e.g. steriods, calcitonin etc.)
* Severe end-organ damage, any malignancy, nephrotic syndrome, malabsorption etc,
* Known case of HIV infection, hyperparathyroidism, granulomatous disorders (e.g. sarcoidosis)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Effects of vitamin D supplementation on structural of atherosclerosis | 2 .5 Years
  Carotid intima media thickness (CIMT) will be measured using a high resolution B-mode ultrasound machine equipped with an 11-MHz frequency linear probe, the procedure will be done by the same radiologist on the same ultrasound machine. All subjects (patients and control) will be examined in supine position, neck extended and chin facing the contralateral side, both common carotid arteries will be examined in both longitudinal and transverse scans, three consecutive measurements of intima media thickness will be taken from the far wall of both common carotid arteries, 1-2 cm proximal to the carotid bulb over the common carotid artery and in the proximal most portion of the internal carotid artery near its origin and the average of these 6 measurements from both sides will taken for final statistical analysis.
Effects of vitamin D supplementation on physiology of atherosclerosis | 2.5 Years
  Brachial artery ultrasound study will be performed in a quiet, dark, temperature-controlled room, all the participants will be in supine position, resting for 10 min, and the measurements of brachial artery will be taken in longitudinal scan in the arm 5-10 cm above the antecubital fossa without permanent vascular access. The luminal diameter of the artery will be measured between the proximal and distal intima.
Effects of vitamin D supplementation on biochemical profile of atherosclerosis | 2.5 Years
  Biochemical: TNF-alpha, hs-CRP, Matrix Metalloproteinase-9.
Effects of vitamin D supplementation on physiology of atherosclerosis | 2.5 Years
  Pulse wave analysis: Using a Mobil-O-Graph (I.E.M., Stolberg, Germany), we will perform pulse wave analyses. The individuals will be performed during the time of pulse wave analysis four BP measurements. The determination of heart rate, peripheral and central pulse pressure, and arterial stiffness of Mobil-O-Graph PWV, also called oPWV, followed all Expert Consensus Document's recommendations on the measurement of Aortic Stiffness 2012.

IPD SHARING:
Plan to Share IPD: No
This study will be conducted at the outpatient department of National Diabetes, Obesity and Cholesterol Foundation (N-DOC), Diabetes Foundation (India) (DFI) and Fortis-C-DOC, Centre of Excellence for Diabetes, Metabolic Diseases and Endocrinology, New Delhi, India.